CLINICAL TRIAL: NCT02168465
Title: Web-Based Self-Management Intervention for Intermittent Urinary Catheter Use
Brief Title: Internet Self-Management for People With Intermittent Urinary Catheters
Acronym: Internet CIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mary Wilde, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5R21NR012763-02 (NIH); 5R21NR012763-02 (NIH)
Record Dates: First submitted 2014-06-17; First posted 2014-06-20 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Spinal Cord Injury
Keywords: self-efficacy; self-management; web-based intervention research
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- teaching self-management of intermittent catheter (Other): Single group pre-post test of feasibility, teaching self-management
  Interventions: Behavioral: teaching self-management of an intermittent catheter

INTERVENTIONS:
Behavioral: teaching self-management of an intermittent catheter — Specifically, we will teach awareness, self-monitoring and self-management strategies to CIC uses with SCI in an online format. Nurse telephone consultation for teaching self-management will be combined with peer leaders for online forums.

SUMMARY:
1. Design and develop web-based self-management intervention to improve catheter-related outcomes and quality of life in people with spinal cord injury (SCI).
2. Conduct a pilot study to assess the feasibility (i.e., acceptability and usability of the website application) and preliminary effectiveness of this new self-management intervention.
3. Develop and test the reliability of new/modified measures (intermittent catheter self-efficacy and self-management).

DETAILED DESCRIPTION:
Stages involve: (1) Develop an Internet-based intervention to improve self-management and outcomes related to clean intermittent catheterization (CIC) among people with SCI (2) Pretest the Internet application with five persons with SCI using CIC; and (3) Conduct a web-based six-month intervention pilot study in a group of 30 with SCI using CIC.

Outcomes are: catheter-related adverse health outcomes (e.g., UTI, urine leakage), CIC self- management, CIC self-efficacy, health related expenditures and quality of life.

Information from this study will be used to modify the Internet application for a future Phase 2 trial in a larger study.

ELIGIBILITY:
Inclusion Criteria:Individuals will be included if they are English speaking adults over 18 years with an SCI and are interested in participating. Inclusion criteria are:

1. use of CIC for regular bladder drainage,
2. expect to use CIC indefinitely or for at least nine months, and
3. access to and ability to use a computer and telephone. Computer and telephone use may be voice activated for those with little hand use. Study participants do not need to perform CIC entirely themselves, as people with limited hand dexterity may have caregivers who do the procedure. They do need to be able to use the computer and telephone however.

Additional inclusion criteria for the five persons in the "intervention and pretesting group" (described below in III, 1) include:

1. having used CIC for regular bladder drainage for at least one year and
2. expect to use CIC indefinitely or for at least one more year. People will need to have used CIC for at least a year so that they are well experienced in CIC because the two Peer Leaders will be selected from this group.

Exclusion Criteria:

* People will be excluded if they cannot communicate in English,
* Are terminally ill, or are expected to discontinue CIC within the next nine months. - Non-English speaking people will not be included because translated instruments (e.g., Spanish) are not available for all measures and doing this as a part of this small study might compromise the integrity of this first test of preliminary effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
catheter-related adverse health outcomes (e.g., UTI, urine leakage) | pre-post 3 month intervention in a single group
  catheter related adverse events will be reported by internet based survey about 3 months after enrollment

SECONDARY OUTCOMES:
Intermittent catheter self-efficacy, | pre-post 3 month intervention in a single group
  Intermittent catheter confidence related to self-care capability

OTHER OUTCOMES:
Intermittent catheter self-management | pre-post 3 month intervention in a single group
  Self-care management involves specific activities performed by the person to manage their intermittent catheter.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States